CLINICAL TRIAL: NCT00658515
Title: A Randomized, Double-blind, Placebo-controlled Study Assessing the Effect of RO4607381 on Cardiovascular Mortality and Morbidity in Clinically Stable Patients With a Recent Acute Coronary Syndrome
Brief Title: A Study of RO4607381 in Stable Coronary Heart Disease Patients With Recent Acute Coronary Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NC20971; 2007-005103-18
Record Dates: First submitted 2008-03-28; First posted 2008-04-15 (Estimated); Results first posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — dalcetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dalcetrapib (RO4607381) (Experimental)
  Interventions: Drug: Dalcetrapib (RO4607381); Drug: Evidence-based medical care for Acute Coronary Syndrome
- Placebo (Placebo Comparator)
  Interventions: Drug: Evidence-based medical care for Acute Coronary Syndrome; Drug: Placebo

INTERVENTIONS:
Drug: Dalcetrapib (RO4607381) — 600mg po daily
  Arms: Dalcetrapib (RO4607381)
Drug: Evidence-based medical care for Acute Coronary Syndrome — As prescribed
Drug: Placebo — po daily
  Arms: Placebo

SUMMARY:
This study will evaluate the potential of RO4607381 to reduce cardiovascular morbidity and mortality in stable coronary heart disease patients with recent Acute Coronary Syndrome (ACS) and evaluate the long term safety profile of the drug. Eligible patients in stable condition will be randomized to receive either RO4607381 600mg po or placebo po, daily, together with a background of standard medication for ACS (including aspirin, antihypertensives and statins). The anticipated time on study treatment is 2+ years, and the target sample size is 15,600 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=45 years of age;
* recently hospitalized for ACS;
* clinically stable;
* receiving evidence-based medical and dietary management of dyslipidemia.

Exclusion Criteria:

* uncontrolled diabetes;
* clinically unstable;
* severe anemia;
* uncontrolled hypertension;
* concomitant treatment with any other drug raising HDL-C (eg niacin, fibrates).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15871 (Actual)
Dates: Start 2008-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (833):
- United States (403):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Tuscaloosa, Alabama
  - Lake Havasu City, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Sierra Vista, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Mountain Home, Arkansas
  - Searcy, Arkansas
  - Anaheim, California
  - Bakersfield, California
  - Bellflower, California
  - Beverly Hills, California
  - Buena Park, California
  - Burbank, California
  - Carmichael, California
  - Corona, California
  - Costa Mesa, California
  - Encinitas, California
  - Fountain Valley, California
  - Fresno, California
  - Fullerton, California
  - Glendale, California
  - Hawaiian Gardens, California
  - Hollywood, California
  - Inglewood, California
  - La Jolla, California
  - La Mesa, California
  - Laguna Hills, California
  - Loma Linda, California
  - Lomita, California
  - Long Beach, California
  - Los Alamitos, California
  - Los Angeles, California
  - Los Banos, California
  - Mather, California
  - Mission Viejo, California
  - Mountain View, California
  - Newport Beach, California
  - Pasadena, California
  - Pomona, California
  - Redondo Beach, California
  - Sacramento, California
  - San Diego, California
  - San Dimas, California
  - San Francisco, California
  - San Jose, California
  - Santa Ana, California
  - Santa Rosa, California
  - Simi Valley, California
  - Stockton, California
  - Thousand Oaks, California
  - Torrance, California
  - Whittier, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Greeley, Colorado
  - Littleton, Colorado
  - Loveland, Colorado
  - Pueblo, Colorado
  - Bridgeport, Connecticut
  - Danbury, Connecticut
  - Guilford, Connecticut
  - Hartford, Connecticut
  - Stamford, Connecticut
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Boynton Beach, Florida
  - Chipley, Florida
  - Clearwater, Florida
  - Crystal River, Florida
  - Daytona Beach, Florida
  - Deerfield Beach, Florida
  - Delray Beach, Florida
  - Elizabeth, Florida
  - Fort Lauderdale, Florida
  - Gainesville, Florida
  - Hollywood, Florida
  - Hudson, Florida
  - Jacksonville, Florida
  - Jacksonville Beach, Florida
  - Jupiter, Florida
  - Kissimmee, Florida
  - Lakeland, Florida
  - Marianna, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Panama City, Florida
  - Pensacola, Florida
  - Plantation, Florida
  - Port Charlotte, Florida
  - Safety Harbor, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Covington, Georgia
  - Decatur, Georgia
  - Monroe, Georgia
  - Riverdale, Georgia
  - Savannah, Georgia
  - Tucker, Georgia
  - Waycross, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Aurora, Illinois
  - Bannockburn, Illinois
  - Chicago, Illinois
  - Evanston, Illinois
  - Gurnee, Illinois
  - Hinsdale, Illinois
  - Joliet, Illinois
  - Libertyville, Illinois
  - Melrose Park, Illinois
  - Mokena, Illinois
  - Naperville, Illinois
  - Normal, Illinois
  - Peoria, Illinois
  - Rockford, Illinois
  - Winfield, Illinois
  - Anderson, Indiana
  - Elkhart, Indiana
  - Evansville, Indiana
  - Fishers, Indiana
  - Fort Wayne, Indiana
  - Franklin, Indiana
  - Greenfield, Indiana
  - Hammond, Indiana
  - Indianapolis, Indiana
  - Merrillville, Indiana
  - Munster, Indiana
  - South Bend, Indiana
  - Ames, Iowa
  - Council Bluffs, Iowa
  - Davenport, Iowa
  - Waterloo, Iowa
  - Olathe, Kansas
  - Overland Park, Kansas
  - Elizabethtown, Kentucky
  - Hazard, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Madisonville, Kentucky
  - Owensboro, Kentucky
  - Alexandria, Louisiana
  - Lake Charles, Louisiana
  - Marrero, Louisiana
  - Metairie, Louisiana
  - Natchitoches, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Slidell, Louisiana
  - West Monroe, Louisiana
  - Bangor, Maine
  - Biddeford, Maine
  - Portland, Maine
  - Scarborough, Maine
  - South Portland, Maine
  - Baltimore, Maryland
  - Bel Air, Maryland
  - Columbia, Maryland
  - Hagerstown, Maryland
  - Pikesville, Maryland
  - Salisbury, Maryland
  - Towson, Maryland
  - Westminster, Maryland
  - Billerica, Massachusetts
  - Boston, Massachusetts
  - East Bridgewater, Massachusetts
  - Haverhill, Massachusetts
  - Hyannis, Massachusetts
  - Natick, Massachusetts
  - North Dartmouth, Massachusetts
  - Pittsfield, Massachusetts
  - Springfield, Massachusetts
  - Taunton, Massachusetts
  - Worcester, Massachusetts
  - Alpena, Michigan
  - Ann Arbor, Michigan
  - Bloomfield, Michigan
  - Cadillac, Michigan
  - Dearborn, Michigan
  - Detroit, Michigan
  - Fairfield, Michigan
  - Flint, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Midland, Michigan
  - Milwaukee, Michigan
  - Petoskey, Michigan
  - Rochester Hills, Michigan
  - Saginaw, Michigan
  - Saint Joseph, Michigan
  - Chaska, Minnesota
  - Duluth, Minnesota
  - Minneapolis, Minnesota
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Saint Cloud, Minnesota
  - Saint Paul, Minnesota
  - Gulfport, Mississippi
  - Jackson, Mississippi
  - Picayune, Mississippi
  - Tupelo, Mississippi
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Great Falls, Montana
  - Kalispell, Montana
  - Missoula, Montana
  - Fremont, Nebraska
  - Grand Island, Nebraska
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Papillion, Nebraska
  - Las Vegas, Nevada
  - Reno, Nevada
  - Manchester, New Hampshire
  - Nashua, New Hampshire
  - Bridgewater, New Jersey
  - Clifton, New Jersey
  - East Orange, New Jersey
  - Edgewater, New Jersey
  - Elmer, New Jersey
  - Greenville, New Jersey
  - Hackensack, New Jersey
  - Haddon Heights, New Jersey
  - Hawthorne, New Jersey
  - Linden, New Jersey
  - Mine Hill, New Jersey
  - New Brunswick, New Jersey
  - Newark, New Jersey
  - Ridgewood, New Jersey
  - Sewell, New Jersey
  - Somerset, New Jersey
  - Summit, New Jersey
  - Toms River, New Jersey
  - Voorhees Township, New Jersey
  - Westwood, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Buffalo, New York
  - Fishkill, New York
  - Flushing, New York
  - Johnson City, New York
  - Liverpool, New York
  - New Hartford, New York
  - New Windsor, New York
  - New York, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Saratoga Springs, New York
  - Springfield Gardens, New York
  - Stony Brook, New York
  - Suffern, New York
  - Syracuse, New York
  - The Bronx, New York
  - Troy, New York
  - West Seneca, New York
  - Asheville, North Carolina
  - Cary, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Concord, North Carolina
  - Durham, North Carolina
  - Elizabeth City, North Carolina
  - Pinehurst, North Carolina
  - Rocky Mount, North Carolina
  - Salt Lake City, North Carolina
  - Tabor City, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Minot, North Dakota
  - Akron, Ohio
  - Athens, Ohio
  - Canton, Ohio
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Kettering, Ohio
  - Mansfield, Ohio
  - Marion, Ohio
  - Mentor, Ohio
  - Middletown, Ohio
  - Sandusky, Ohio
  - Springfield, Ohio
  - Thornville, Ohio
  - Toledo, Ohio
  - Westlake, Ohio
  - Willoughby Hills, Ohio
  - Zanesville, Ohio
  - Bartlesville, Oklahoma
  - Midwest City, Oklahoma
  - Oklahoma City, Oklahoma
  - Bend, Oregon
  - Portland, Oregon
  - Abington, Pennsylvania
  - Allentown, Pennsylvania
  - Altoona, Pennsylvania
  - Beaver, Pennsylvania
  - Bryn Mawr, Pennsylvania
  - Camp Hill, Pennsylvania
  - Downingtown, Pennsylvania
  - Doylestown, Pennsylvania
  - Easton, Pennsylvania
  - Erie, Pennsylvania
  - Feasterville, Pennsylvania
  - Havertown, Pennsylvania
  - Hershey, Pennsylvania
  - Lancaster, Pennsylvania
  - Langhorne, Pennsylvania
  - Limerick, Pennsylvania
  - Natrona Heights, Pennsylvania
  - North Wales, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Pottstown, Pennsylvania
  - Sayre, Pennsylvania
  - Scranton, Pennsylvania
  - Sellersville, Pennsylvania
  - West Chester, Pennsylvania
  - Wormleysburg, Pennsylvania
  - Wynnewood, Pennsylvania
  - Wyomissing, Pennsylvania
  - Providence, Rhode Island
  - Wakefield, Rhode Island
  - Aiken, South Carolina
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greer, South Carolina
  - Moncks Corner, South Carolina
  - Spartanburg, South Carolina
  - Taylors, South Carolina
  - Knoxville, South Dakota
  - Rapid City, South Dakota
  - Sioux Falls, South Dakota
  - Bristol, Tennessee
  - Jackson, Tennessee
  - Johnson City, Tennessee
  - Kingsport, Tennessee
  - Knoxville, Tennessee
  - Lexington, Tennessee
  - Oak Ridge, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Humble, Texas
  - Killeen, Texas
  - Lubbock, Texas
  - Odessa, Texas
  - Plano, Texas
  - Round Rock, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Tyler, Texas
  - Victoria, Texas
  - Layton, Utah
  - Provo, Utah
  - Burke, Virginia
  - Charlottesville, Virginia
  - Colonial Heights, Virginia
  - Danville, Virginia
  - Falls Church, Virginia
  - Galax, Virginia
  - Hopewell, Virginia
  - Manassas, Virginia
  - Midlothian, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Roanoke, Virginia
  - Salem, Virginia
  - Springfield, Virginia
  - Winchester, Virginia
  - Bellevue, Washington
  - Everett, Washington
  - Monroe, Washington
  - Selah, Washington
  - Spokane, Washington
  - Clarksburg, West Virginia
  - Beloit, Wisconsin
  - Burlington, Wisconsin
  - Green Bay, Wisconsin
  - La Crosse, Wisconsin
  - Madison, Wisconsin
  - Marshfield, Wisconsin
  - Milwaukee, Wisconsin
- Argentina (24):
  - Almirante Brown
  - Bahía Blanca
  - Buenos Aires
  - CABA
  - Capital Federal
  - Cipolletti
  - Ciudad Autonoma Bs As
  - Ciudad Autónoma de Bs. As.
  - Coronel Suárez
  - Corrientes
  - Córdoba
  - Junín
  - La Plata
  - Mar del Plata
  - Mendoza
  - Quilmes
  - Rosario
  - Salta
  - San Isidro
  - San Justo
  - San Martín
  - San Miguel de Tucumán
  - San Salvador de Jujuy
  - Santa Fe
- Australia (16):
  - Garran, Australian Capital Territory
  - Coffs Harbour, New South Wales
  - Concord, New South Wales
  - Epping, New South Wales
  - Kingswood, New South Wales
  - Wollongong, New South Wales
  - Cairns, Queensland
  - Chermside, Queensland
  - Milton, Queensland
  - Woolloongabba, Queensland
  - Bedford Park, South Australia
  - Box Hill, Victoria
  - Geelong, Victoria
  - Sale, Victoria
  - Joondalup, Western Australia
  - Nedlands, Western Australia
- Austria (4):
  - Feldkirch
  - Graz
  - Linz
  - Vienna
- Belgium (8):
  - Aalst
  - Bruges
  - Brussels
  - Genk
  - Ghent
  - La Louvière
  - Roeselare
  - Tienen
- Brazil (22):
  - Maceió, Alagoas
  - Fortaleza, Ceará
  - Salvador, Estado de Bahia
  - Goiânia, Goiás
  - Campo Grande, Mato Grosso do Sul
  - Belo Horizonte, Minas Gerais
  - Uberlândia, Minas Gerais
  - Campina Grande do Sul, Paraná
  - Curitiba, Paraná
  - Olinda, Pernambuco
  - Recife, Pernambuco
  - Rio de Janeiro, Rio de Janeiro
  - Natal, Rio Grande do Norte
  - Pelotas, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Sao Jose Do Rio Preto, Santa Catarina
  - Aracaju, Sergipe
  - Campinas, São Paulo
  - Ribeirão Preto, São Paulo
  - Santo André, São Paulo
  - São José do Rio Preto, São Paulo
  - São Paulo, São Paulo
- Canada (46):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Nanaimo, British Columbia
  - New Westminster, British Columbia
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - Mount Pearl, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Ajax, Ontario
  - Brampton, Ontario
  - Burlington, Ontario
  - Cambridge, Ontario
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Kingston, Ontario
  - Kitchener, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Gatineau, Quebec
  - Granby, Quebec
  - Greenfield Park, Quebec
  - Lachine, Quebec
  - Laval, Quebec
  - Longueuil, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint Georges-de-beauce, Quebec
  - Saint-Charles-Borromée, Quebec
  - Saint-Jérôme, Quebec
  - Saint-Lambert, Quebec
  - Saint-Léonard, Quebec
  - Sherbrooke, Quebec
  - Ste. Foy, Quebec
  - Terrebonne, Quebec
  - Trois-Rivières, Quebec
  - Val-d'Or, Quebec
  - Westmount, Quebec
  - Saskatoon, Saskatchewan
- China (18):
  - Beijing
  - Changsha
  - Dalian
  - Daqing
  - Guangzhou
  - Hangzhou
  - Harbin
  - Jinan
  - Lanzhou
  - Nanchang
  - Nanjing
  - Shanghai
  - Shenyang
  - Shijiazhuang
  - Suzhou
  - Wenzhou
  - Wuhan
  - Xi'an
- Czechia (19):
  - Brno
  - Chrudim
  - České Budějovice
  - Hradec Králové
  - Jihlava
  - Jindřichův Hradec
  - Karlovy Vary
  - Kroměříž
  - Náchod
  - Ostrava - Fifejdy
  - Pardubice
  - Prague
  - Semily
  - Slaný
  - Tábor
  - Teplice
  - Trutnov
  - Zlín
  - Znojmo
- Denmark (10):
  - Frederiksberg
  - Hellerup
  - Herlev
  - Herning
  - Hillerød
  - Kolding
  - København S
  - Køge
  - Roskilde
  - Svendborg
- Finland (3):
  - Jyväskylä
  - Kotka
  - Kuopio
- France (16):
  - Angers
  - Bron
  - Colmar
  - Dijon
  - Lille
  - Marseille
  - Montfermeil
  - Paris
  - Pessac
  - Poitiers
  - Roubaix
  - Saint-Herblain
  - Strasbourg
  - Tourcoing
  - Valenciennes
  - Vandœuvre-lès-Nancy
- Germany (31):
  - Bad Krozingen
  - Bad Rothenfelde
  - Bad Segeberg
  - Berlin
  - Bielefeld
  - Bochum
  - Burg
  - Coburg
  - Darmstadt
  - Dortmund
  - Duisburg
  - Essen
  - Frankfurt
  - Frankfurt am Main
  - Führt
  - Halle
  - Hamburg
  - Heidelberg
  - Homburg/Saar
  - Langen
  - Limburg
  - Mainz
  - Mannheim
  - Mönchengladbach
  - Neuss
  - Northeim
  - Rüdersdorf
  - Ulm
  - Villingen-Schwenningen
  - Witten
  - Wuppertal
- Toulouse, Grenada
- Hungary (12):
  - Baja
  - Békéscsaba
  - Budapest
  - Debrecen
  - Kalocsa
  - Kecskemét
  - Pécs
  - Sopron
  - Szeged
  - Szekszárd
  - Székesfehérvár
  - Zalaegerszeg
- Dublin, Ireland
- Israel (15):
  - Afula
  - Beersheba
  - Giv‘atayim
  - Hadera
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Nazareth
  - Petah Tikva
  - Rehovot
  - Tel Aviv
  - Tel Litwinsky
  - Tiberias
  - Ẕerifin
- Italy (21):
  - Chieti, Abruzzo
  - Caserta, Campania
  - Napoli, Campania
  - Carpi, Emilia-Romagna
  - Forlì, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Piacenza, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Genoa, Liguria
  - Bergamo, Lombardy
  - Como, Lombardy
  - Milan, Lombardy
  - Pavia, Lombardy
  - Rozzano, Lombardy
  - Novara, Piedmont
  - Turin, Piedmont
  - Pesaro, The Marches
  - Castelnuovo, Tuscany
  - S. Bonifacio, Veneto
  - Treviso, Veneto
- Netherlands (37):
  - 's-Hertogenbosch
  - Alkmaar
  - Almelo
  - Amersfoort
  - Amstelveen
  - Amsterdam
  - Arnhem
  - Blaricum
  - Breda
  - Capelle AD Yssel
  - Delft
  - Den Helder
  - Deventer
  - Eindhoven
  - Enschede
  - Goes
  - Groningen
  - Haarlem
  - Heerlen
  - Hengelo
  - Hilversum
  - Hoofddorp
  - Hoorn
  - Leiden
  - Leiderdorp
  - Maastricht
  - Nieuwegein
  - Nijmegen
  - Purmerend
  - Rotterdam
  - Sneek
  - Stadskanaal
  - Tilburg
  - Utrecht
  - Weert
  - Zaandam
  - Zwolle
- New Zealand (7):
  - Auckland
  - Christchurch
  - Dunedin
  - Hamilton
  - Nelson
  - New Plymouth
  - Wellington
- Poland (30):
  - Bialystok
  - Bydgoszcz
  - Elblag
  - Gdansk
  - Gdynia
  - Grodzisk Mazowiecki
  - Inowrocław
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Nowa Sól
  - Poznan
  - Puławy
  - Płock
  - Ruda Śląska
  - Siedlce
  - Sopot
  - Sosnowiec
  - Stalowa Wola
  - Starachowice
  - Szczecin
  - Świdnik
  - Tarnów
  - Torun
  - Warsaw
  - Wałbrzych
  - Wroclaw
  - Zamość
  - Zielona Góra
- Puerto Rico (7):
  - Aguas Buenas
  - Caguas
  - Manatí
  - Ponce
  - Río Grande
  - San Juan
  - Toa Baja
- Slovakia (8):
  - Banská Bystrica
  - Bardejov
  - Bratislava
  - Dolný Kubín
  - Martin
  - Nitra
  - Rimavská Sobota
  - Žilina
- South Africa (11):
  - Alberton
  - Bloemfontein
  - Boksburg
  - Durban
  - Johannesburg
  - Kuilsriver
  - Lyttelton, Pretoria
  - Panorama
  - Pinelands
  - Pretoria
  - Somerset West
- South Korea (9):
  - Busan
  - Daegu
  - Gangwon-Do
  - Gangwon-do
  - Gwangju
  - Gyeonggi-do
  - Incheon
  - Kyonggi-do
  - Seoul
- Spain (20):
  - Vitoria-Gasteiz, Alava
  - Sant Joan d'Alacant, Alicante
  - L'Hospitalet de Llobregat, Barcelona
  - Santander, Cantabria
  - Figueres, Girona
  - Santiago de Compostela, LA Coruña
  - Majadahonda, Madrid
  - Málaga, Malaga
  - Pamplona, Navarre
  - Vigo, Pontevedra
  - Seville, Sevilla
  - Alicante
  - Almería
  - Barcelona
  - Guadalajara
  - Lugo
  - Madrid
  - Tarragona
  - Valencia
  - Valladolid
- Sweden (4):
  - Falun
  - Gothenburg
  - Stockholm
  - Västerås
- Switzerland (7):
  - Fribourg
  - Geneva
  - Kreuzlingen
  - Lucerne
  - Lugano
  - Münsterlingen
  - Wolhusen
- United Kingdom (23):
  - Airdrie
  - Barnet
  - Belfast
  - Birmingham
  - Blackpool
  - Bradford
  - Cambridge
  - Chertsey
  - Edinburgh
  - Glasgow
  - Larbert
  - Leicester
  - London
  - Luton
  - Manchester
  - Middlesbrough
  - Middlesex
  - Nottingham
  - Nuneaton
  - Paisley
  - Peterborough
  - Stockport
  - Swansea

REFERENCES:
- [Derived] Schwartz GG, Leiter LA, Ballantyne CM, Barter PJ, Black DM, Kallend D, Laghrissi-Thode F, Leitersdorf E, McMurray JJV, Nicholls SJ, Olsson AG, Preiss D, Shah PK, Tardif JC, Kittelson J. Dalcetrapib Reduces Risk of New-Onset Diabetes in Patients With Coronary Heart Disease. Diabetes Care. 2020 May;43(5):1077-1084. doi: 10.2337/dc19-2204. Epub 2020 Mar 6. PMID 32144166
- [Derived] Salahuddin T, Kittelson J, Tardif JC, Shah PK, Olsson AG, Nicholls SJ, Leitersdorf E, Leiter LA, Kallend D, Black DM, Barter PJ, Ballantyne CM, Schwartz GG. Association of high-density lipoprotein particle concentration with cardiovascular risk following acute coronary syndrome: A case-cohort analysis of the dal-Outcomes trial. Am Heart J. 2020 Mar;221:60-66. doi: 10.1016/j.ahj.2019.12.003. Epub 2019 Dec 16. PMID 31927126
- [Derived] Schwartz GG, Ballantyne CM, Barter PJ, Kallend D, Leiter LA, Leitersdorf E, McMurray JJV, Nicholls SJ, Olsson AG, Shah PK, Tardif JC, Kittelson J. Association of Lipoprotein(a) With Risk of Recurrent Ischemic Events Following Acute Coronary Syndrome: Analysis of the dal-Outcomes Randomized Clinical Trial. JAMA Cardiol. 2018 Feb 1;3(2):164-168. doi: 10.1001/jamacardio.2017.3833. PMID 29071331
- [Derived] Pitts R, Gunzburger E, Ballantyne CM, Barter PJ, Kallend D, Leiter LA, Leitersdorf E, Nicholls SJ, Shah PK, Tardif JC, Olsson AG, McMurray JJ, Kittelson J, Schwartz GG. Aldosterone Does Not Predict Cardiovascular Events Following Acute Coronary Syndrome in Patients Initially Without Heart Failure. J Am Heart Assoc. 2017 Jan 10;6(1):e004119. doi: 10.1161/JAHA.116.004119. PMID 28073769
- [Derived] Tardif JC, Rhainds D, Brodeur M, Feroz Zada Y, Fouodjio R, Provost S, Boule M, Alem S, Gregoire JC, L'Allier PL, Ibrahim R, Guertin MC, Mongrain I, Olsson AG, Schwartz GG, Rheaume E, Dube MP. Genotype-Dependent Effects of Dalcetrapib on Cholesterol Efflux and Inflammation: Concordance With Clinical Outcomes. Circ Cardiovasc Genet. 2016 Aug;9(4):340-8. doi: 10.1161/CIRCGENETICS.116.001405. Epub 2016 Jul 14. PMID 27418594
- [Derived] Schwartz GG, Abt M, Bao W, DeMicco D, Kallend D, Miller M, Mundl H, Olsson AG. Fasting triglycerides predict recurrent ischemic events in patients with acute coronary syndrome treated with statins. J Am Coll Cardiol. 2015 Jun 2;65(21):2267-75. doi: 10.1016/j.jacc.2015.03.544. PMID 26022813
- [Derived] Tardif JC, Rheaume E, Lemieux Perreault LP, Gregoire JC, Feroz Zada Y, Asselin G, Provost S, Barhdadi A, Rhainds D, L'Allier PL, Ibrahim R, Upmanyu R, Niesor EJ, Benghozi R, Suchankova G, Laghrissi-Thode F, Guertin MC, Olsson AG, Mongrain I, Schwartz GG, Dube MP. Pharmacogenomic determinants of the cardiovascular effects of dalcetrapib. Circ Cardiovasc Genet. 2015 Apr;8(2):372-82. doi: 10.1161/CIRCGENETICS.114.000663. Epub 2015 Jan 11. PMID 25583994
- [Derived] Schwartz GG, Olsson AG, Abt M, Ballantyne CM, Barter PJ, Brumm J, Chaitman BR, Holme IM, Kallend D, Leiter LA, Leitersdorf E, McMurray JJ, Mundl H, Nicholls SJ, Shah PK, Tardif JC, Wright RS; dal-OUTCOMES Investigators. Effects of dalcetrapib in patients with a recent acute coronary syndrome. N Engl J Med. 2012 Nov 29;367(22):2089-99. doi: 10.1056/NEJMoa1206797. Epub 2012 Nov 5. PMID 23126252
- [Derived] Luscher TF, Taddei S, Kaski JC, Jukema JW, Kallend D, Munzel T, Kastelein JJ, Deanfield JE; dal-VESSEL Investigators. Vascular effects and safety of dalcetrapib in patients with or at risk of coronary heart disease: the dal-VESSEL randomized clinical trial. Eur Heart J. 2012 Apr;33(7):857-65. doi: 10.1093/eurheartj/ehs019. Epub 2012 Feb 16. PMID 22345126
- [Derived] Derks M, Abt M, Parr G, Meneses-Lorente G, Young AM, Phelan M. No clinically relevant drug-drug interactions when dalcetrapib is co-administered with atorvastatin. Expert Opin Investig Drugs. 2010 Oct;19(10):1135-45. doi: 10.1517/13543784.2010.509342. PMID 20738227
- [Derived] Schwartz GG, Olsson AG, Ballantyne CM, Barter PJ, Holme IM, Kallend D, Leiter LA, Leitersdorf E, McMurray JJ, Shah PK, Tardif JC, Chaitman BR, Duttlinger-Maddux R, Mathieson J; dal-OUTCOMES Committees and Investigators. Rationale and design of the dal-OUTCOMES trial: efficacy and safety of dalcetrapib in patients with recent acute coronary syndrome. Am Heart J. 2009 Dec;158(6):896-901.e3. doi: 10.1016/j.ahj.2009.09.017. PMID 19958854
- [Derived] Stein EA, Stroes ES, Steiner G, Buckley BM, Capponi AM, Burgess T, Niesor EJ, Kallend D, Kastelein JJ. Safety and tolerability of dalcetrapib. Am J Cardiol. 2009 Jul 1;104(1):82-91. doi: 10.1016/j.amjcard.2009.02.061. PMID 19576325

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Started | 7938 | 7933
Completed | 7626 | 7668
Not Completed | 312 | 265

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalcetrapib (RO4607381) | Placebo | Total
Number analyzed (Participants) | 7938 | 7933 | 15871
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (9.09) | 60.1 (9.10) | 60.2 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6365 | 6436 | 12801
  Male | 1573 | 1497 | 3070

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Cardiovascular Mortality and Morbidity
Description: Number of cardiovascular events per patient per year
Time Frame: From date of randomization to first event up to 48 months
Measure: Number; unit: Event per Patient Years of Followup
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 7938 | 7933
Event per Patient Years of Followup | 0.034050 | 0.032759

2. Secondary Outcome: Composite Endpoint:All Cause Mortality
Time Frame: Throughout Study, up to 53 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 7938 | 7933
Participants | 226 | 229

3. Secondary Outcome: Change From Baseline for HDL Cholesterol
Time Frame: At 53 Months
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 7938 | 7933
mg/dL | 44.96 (4.133) | 15.60 (4.102)

4. Secondary Outcome: Adverse Events, Lab Parameters, Vital Signs, ECG
Time Frame: Throughout Study, up to 53 Months
Population: Data not collected
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Serious Adverse Events (participants affected / at risk) | 1688/7938 | 1692/7933
Other Adverse Events (participants affected / at risk) | 4487/7938 | 4297/7933
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalcetrapib (RO4607381) (N=7938) | Placebo (N=7933)
Angina Pectoris (Cardiac disorders) | 114 | 116
Atrial Fibrillation (Cardiac disorders) | 69 | 77
Angina Unstable (Cardiac disorders) | 49 | 39
Ventricular Tachycardia (Cardiac disorders) | 18 | 16
Atrial Flutter (Cardiac disorders) | 7 | 13
Coronary Artery Disease (Cardiac disorders) | 11 | 8
Sick Sinus Syndrome (Cardiac disorders) | 8 | 10
Bradycardia (Cardiac disorders) | 6 | 8
Ischemia Cardiomyopathy (Cardiac disorders) | 8 | 5
Aortic Valve Stenosis (Cardiac disorders) | 5 | 5
Palpitations (Cardiac disorders) | 4 | 6
Arrhythmia (Cardiac disorders) | 4 | 5
Atrioventricular Block Complete (Cardiac disorders) | 5 | 4
Myocardial Ischemia (Cardiac disorders) | 5 | 4
Supraventricular Tachycardia (Cardiac disorders) | 5 | 4
Ventricular Extrasystole (Cardiac disorders) | 3 | 5
Mitral Valve Incomplete (Cardiac disorders) | 5 | 2
Atrial Tachicardia (Cardiac disorders) | 4 | 1
Atrioventricular Block Second Degreee (Cardiac disorders) | 1 | 4
Cariogenic Shock (Cardiac disorders) | 2 | 3
Pericardial Effusion (Cardiac disorders) | 2 | 2
Prinzmetal Angina (Cardiac disorders) | 2 | 2
Sinus Bradycardia (Cardiac disorders) | 2 | 2
Sinus Tachycardia (Cardiac disorders) | 3 | 1
Tachyarrhythmia (Cardiac disorders) | 2 | 2
Tachycardia (Cardiac disorders) | 2 | 2
Bradyarrhythmia (Cardiac disorders) | 2 | 1
Dressler's Syndrome (Cardiac disorders) | 1 | 2
Left Ventricular Dysfunction (Cardiac disorders) | 2 | 1
Pericarditis (Cardiac disorders) | 1 | 2
Aortic Valve Incompetence (Cardiac disorders) | 1 | 1
Arteriospasm Coronary (Cardiac disorders) | 2 | 0
Cardiac Discomfort (Cardiac disorders) | 0 | 2
Cardiac Tamponade (Cardiac disorders) | 1 | 1
Intracardiac Thrombus (Cardiac disorders) | 1 | 1
Rhythm Idioventricular (Cardiac disorders) | 0 | 2
Sinus Arrest (Cardiac disorders) | 0 | 2
Sinus Arrhythmia (Cardiac disorders) | 1 | 1
Ventricular Hypokinesia (Cardiac disorders) | 1 | 1
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Aortic Valve Disease (Cardiac disorders) | 0 | 1
Aortic Valve Disease Mixed (Cardiac disorders) | 1 | 0
Arrhythmia Supraventricular (Cardiac disorders) | 1 | 0
Brugada Syndrome (Cardiac disorders) | 1 | 0
Bundle Branch Block Right (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Asthma (Cardiac disorders) | 0 | 1
Cardiac Disorder (Cardiac disorders) | 0 | 1
Cardiac Pseudoaneurism (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Conduction Disorder (Cardiac disorders) | 1 | 0
Coronary Artery Dissection (Cardiac disorders) | 0 | 1
Coronary Artery Insufficiency (Cardiac disorders) | 1 | 0
Long QT Syndrome (Cardiac disorders) | 0 | 1
Mitral Valve Disease (Cardiac disorders) | 1 | 0
Mitral Valve Prolapse (Cardiac disorders) | 0 | 1
Pericardial Hemorrhage (Cardiac disorders) | 1 | 0
Tricuspid Valve Incompetence (Cardiac disorders) | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 0 | 1
Ventricular Fibrillation (Cardiac disorders) | 0 | 1
Ventricular Tachyarrhythmia (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 64 | 72
Cellulitis (Infections and infestations) | 22 | 22
Appendicitis (Infections and infestations) | 14 | 20
Urinary Tract Infection (Infections and infestations) | 12 | 21
Gastroenteritis (Infections and infestations) | 13 | 12
Diverticulitis (Infections and infestations) | 10 | 11
Bronchitis (Infections and infestations) | 7 | 12
Erysipelas (Infections and infestations) | 3 | 10
Sepsis (Infections and infestations) | 8 | 4
Urosepsis (Infections and infestations) | 5 | 6
Wound Infection (Infections and infestations) | 3 | 6
Septic Shock (Infections and infestations) | 2 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 3
Appendicitis Perforated (Infections and infestations) | 3 | 4
Bronchopneumonia (Infections and infestations) | 5 | 2
Herpes Zoster (Infections and infestations) | 2 | 5
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 4 | 3
Respiratory Tract Infection (Infections and infestations) | 3 | 4
Viral Infection (Infections and infestations) | 1 | 6
Anal Abscess (Infections and infestations) | 3 | 3
Gangrene (Infections and infestations) | 3 | 3
Lower Respiratory Tract Infection (Infections and infestations) | 5 | 1
Lung Infection (Infections and infestations) | 2 | 4
Osteomyelitis (Infections and infestations) | 1 | 5
Pyelonephritis (Infections and infestations) | 3 | 3
Sinusitis (Infections and infestations) | 2 | 3
Staphylococcal Infections (Infections and infestations) | 0 | 5
Vestibular Neuronitis (Infections and infestations) | 3 | 2
Hepatitis B (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 1 | 3
Pyelonephritis Acute (Infections and infestations) | 2 | 2
Abdominal Abscess (Infections and infestations) | 2 | 1
Bursitis Infective (Infections and infestations) | 2 | 1
Device Related Infection (Infections and infestations) | 1 | 2
Endocarditis (Infections and infestations) | 1 | 2
Escherichia Urinary Tract Infection (Infections and infestations) | 3 | 0
Gastroenteritis Viral (Infections and infestations) | 3 | 0
Hematoma Infection (Infections and infestations) | 1 | 2
Helicobacter Gastritis (Infections and infestations) | 2 | 1
Localized Injection (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 1 | 2
Pneumonia Bacterial (Infections and infestations) | 1 | 2
Pneumonia Primary Atypical (Infections and infestations) | 3 | 0
Skin Infection (Infections and infestations) | 2 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Campylobacter Gastroenteritis (Infections and infestations) | 0 | 2
Chronic Sinusitis (Infections and infestations) | 1 | 1
Clostridium Difficile Sepsis (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 1 | 1
Diarrhea Infectious (Infections and infestations) | 1 | 1
Enterocolitis Infectious (Infections and infestations) | 0 | 2
Gastroenteritis Salmonella (Infections and infestations) | 0 | 2
Groin Abscess (Infections and infestations) | 1 | 1
Incision Site Infection (Infections and infestations) | 0 | 2
Infected Skin Ulcer (Infections and infestations) | 2 | 0
Joint Abscess (Infections and infestations) | 2 | 0
Liver Abscess (Infections and infestations) | 2 | 0
Otitis Media Chronic (Infections and infestations) | 2 | 0
Perirectal Abscess (Infections and infestations) | 1 | 1
Post Procedural Sepsis (Infections and infestations) | 1 | 1
Postoperative Wound Infection (Infections and infestations) | 2 | 0
Pulmonary Sepsis (Infections and infestations) | 1 | 1
Scrotal Abscess (Infections and infestations) | 1 | 1
Sialoadenitis (Infections and infestations) | 1 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 2 | 0
Tracheobronchitis (Infections and infestations) | 0 | 2
Wound Abscess (Infections and infestations) | 0 | 2
Wound Infection Staphylococcal (Infections and infestations) | 0 | 2
Abdominal Sepsis (Infections and infestations) | 0 | 1
Abdominal Wall Abscess (Infections and infestations) | 0 | 1
Abdominal Wall Infection (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Abscess Neck (Infections and infestations) | 0 | 1
Acute Tonsillitis (Infections and infestations) | 0 | 1
Appendiceal Abscess (Infections and infestations) | 1 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 1
Arthritis Infective (Infections and infestations) | 0 | 1
Aspergillosis (Infections and infestations) | 1 | 0
Blister Infected (Infections and infestations) | 0 | 1
Bronchitis Viral (Infections and infestations) | 1 | 0
Campylobacter Infection (Infections and infestations) | 0 | 1
Cellulitis of External Male Genital Organ (Infections and infestations) | 1 | 0
Cellulitis Orbital (Infections and infestations) | 0 | 1
Cellulitis Staphylococcus (Infections and infestations) | 1 | 0
Clostridial Infection (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Coccidioidomycosis (Infections and infestations) | 1 | 0
Dengue Fever (Infections and infestations) | 0 | 1
Diabetic Foot Infection (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia Sepsis (Infections and infestations) | 1 | 0
Extradural Abscess (Infections and infestations) | 0 | 1
Febrile Infection (Infections and infestations) | 1 | 0
Gastric Ulcer Helicobacter (Infections and infestations) | 0 | 1
Giardiasis (Infections and infestations) | 0 | 1
Haemophilus Infection (Infections and infestations) | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 1
Herpes Zoster Ophthalmic (Infections and infestations) | 1 | 0
Infected Dermal Cyst (Infections and infestations) | 1 | 0
Injection Site Cellulitis (Infections and infestations) | 0 | 1
Klebsiella Sepsis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0
Mediastinitis (Infections and infestations) | 0 | 1
Meningitis Herpes (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Parotid Abscess (Infections and infestations) | 0 | 1
Peridiverticular Abscess (Infections and infestations) | 1 | 0
Peritoneal Abscess (Infections and infestations) | 1 | 0
Peritonsillar Abscess (Infections and infestations) | 1 | 0
Pharyngeal Abscess (Infections and infestations) | 1 | 0
Pleurisy Viral (Infections and infestations) | 1 | 0
Pneumococcal Infection (Infections and infestations) | 1 | 0
Pneumonia Influenzal (Infections and infestations) | 0 | 1
Pneumonia Legionella (Infections and infestations) | 0 | 1
Pneumonia Viral (Infections and infestations) | 1 | 0
Post Procedural Infection (Infections and infestations) | 1 | 0
Postoperative Abscess (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Rectal Abscess (Infections and infestations) | 1 | 0
Respiratory Moniliasis (Infections and infestations) | 1 | 0
Scrub Typhus (Infections and infestations) | 1 | 0
Septic Encephalopathy (Infections and infestations) | 0 | 1
Soft Tissue Infection (Infections and infestations) | 0 | 1
Staphylococcal Abscess (Infections and infestations) | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 1
Staphylococcal Skin Infection (Infections and infestations) | 0 | 1
Streptococcal Bacteremia (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Tracheostomy Infection (Infections and infestations) | 1 | 0
Viral Myocarditis (Infections and infestations) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 145 | 152
Chest Pain (General disorders) | 97 | 103
Chest Discomfort (General disorders) | 12 | 14
Pyrexia (General disorders) | 3 | 4
Asthenia (General disorders) | 1 | 4
Edema Peripheral (General disorders) | 3 | 1
Multi-Organ Failure (General disorders) | 2 | 1
Device Dislocation (General disorders) | 1 | 1
Device Malfunction (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 2
Pain (General disorders) | 0 | 2
Spinal Pain (General disorders) | 1 | 1
Catheter Site Hematoma (General disorders) | 0 | 1
Chronic Fatigue Syndrome (General disorders) | 0 | 1
Device Damage (General disorders) | 0 | 1
Drug Intolerance (General disorders) | 1 | 0
Gait Disturbance (General disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 1 | 0
Granuloma (General disorders) | 0 | 1
Hernia (General disorders) | 0 | 1
Hernia Obstructive (General disorders) | 0 | 1
Impaired Healing (General disorders) | 1 | 0
Implant Site Inflammation (General disorders) | 0 | 1
Local Swelling (General disorders) | 1 | 0
Polyserositis (General disorders) | 1 | 0
Pseudocyst (General disorders) | 0 | 1
Puncture Site Hemorrhage (General disorders) | 1 | 0
Soft Tissue Inflammation (General disorders) | 0 | 1
Vessel Puncture Site Hematoma (General disorders) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 31 | 34
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 15
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 11
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 8
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 11
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 8
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 6
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 5
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 8
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 2
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Lung Squamous Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Benign Neoplasm of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Chronic Lymphocytic Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Renal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Acute Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lip And/Or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Melodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Non-Hodgkins Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Esophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Acute Monocytic Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast Cancer In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Meningioma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metasteses To Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic Carcinoid Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Esophageal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Parathyroid Tumor Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pituitary Tumor Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basosquamous Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign Gastric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Biliary Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Adenocarcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Papiloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Squamous Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Transitional Cell Carcinoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Burkit's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid Tumor Of The Gastrointestinal Tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoma Tumor Of The Small Bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic Myolomonocytic Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer Stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Extranodal Marginal Zone B-Cell Lymphoma (Malt Type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal Stromal Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Inflammatory Pseudotumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal Papilloma Of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal Cancer Stage 0 Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lentigo Maligna Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Adenocarcinoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Adenocarcinoma Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Fibrous Histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metasteses To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic Uterine Cancer Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Esophageal Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Epithelial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paget's Disease Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sebaceous Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spindle Cell Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thymoma Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumor Perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 14 | 21
Inguinal Hernia (Gastrointestinal disorders) | 13 | 17
Abdominal Pain (Gastrointestinal disorders) | 11 | 15
Gastritis (Gastrointestinal disorders) | 8 | 10
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 8 | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 7 | 9
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 11 | 5
Small Intestinal Obstruction (Gastrointestinal disorders) | 11 | 5
Diarrhea (Gastrointestinal disorders) | 7 | 7
Pancreatitis (Gastrointestinal disorders) | 7 | 7
Pancreatitis Acute (Gastrointestinal disorders) | 8 | 6
Dyspepsia (Gastrointestinal disorders) | 7 | 6
Gastric Ulcer Hemorrhage (Gastrointestinal disorders) | 2 | 9
Colonic Polyp (Gastrointestinal disorders) | 4 | 6
Duodenal Ulcer Hemorrhage (Gastrointestinal disorders) | 6 | 4
Gastric Ulcer (Gastrointestinal disorders) | 5 | 5
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 7 | 1
Constipation (Gastrointestinal disorders) | 3 | 4
Rectal Hemorrhage (Gastrointestinal disorders) | 6 | 1
Diverticular Perforation (Gastrointestinal disorders) | 1 | 4
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 5
Gastric Hemorrhage (Gastrointestinal disorders) | 2 | 3
Ileus (Gastrointestinal disorders) | 3 | 2
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 4 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 4 | 0
Colitis (Gastrointestinal disorders) | 2 | 2
Diverticulum Intestinal Hemorrhagic (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 3
Hematemesis (Gastrointestinal disorders) | 1 | 3
Hemorrhoids (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 3
Esophagitis (Gastrointestinal disorders) | 3 | 1
Diverticulitis Intestinal Hemorrhagic (Gastrointestinal disorders) | 1 | 2
Diverticulum (Gastrointestinal disorders) | 3 | 0
Diverticulum Intestinal (Gastrointestinal disorders) | 3 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 2
Gastritis Erosive (Gastrointestinal disorders) | 1 | 2
Gastritis Hemorrhagic (Gastrointestinal disorders) | 3 | 0
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 2 | 1
Esophageal Hemorrhage (Gastrointestinal disorders) | 2 | 1
Umbilical Hernia (Gastrointestinal disorders) | 2 | 1
Abdominal Hernia (Gastrointestinal disorders) | 1 | 1
Appendix Disorder (Gastrointestinal disorders) | 1 | 1
Barrett's Esophagus (Gastrointestinal disorders) | 1 | 1
Colitis Ischemic (Gastrointestinal disorders) | 1 | 1
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 2
Crohn's Disease (Gastrointestinal disorders) | 0 | 2
Duodenitis (Gastrointestinal disorders) | 1 | 1
Gastroduodenal Ulcer (Gastrointestinal disorders) | 1 | 1
Gastroesophagitis (Gastrointestinal disorders) | 1 | 1
Hematochezia (Gastrointestinal disorders) | 2 | 0
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1 | 1
Intestinal Hemorrhage (Gastrointestinal disorders) | 2 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2
Intestinal Perforation (Gastrointestinal disorders) | 1 | 1
Large Intestinal Ulcer Hemorrhage (Gastrointestinal disorders) | 0 | 2
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Esophageal Stenosis (Gastrointestinal disorders) | 0 | 2
Esophageal Ulcer Hemorrhage (Gastrointestinal disorders) | 1 | 1
Peptic Ulcer (Gastrointestinal disorders) | 0 | 2
Peptic Ulcer Hemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal Distention (Gastrointestinal disorders) | 0 | 1
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0
Abdominal Wall Hematoma (Gastrointestinal disorders) | 0 | 1
Acute Abdomen (Gastrointestinal disorders) | 1 | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 1
Anal Fistula (Gastrointestinal disorders) | 1 | 0
Colitis Microscopic (Gastrointestinal disorders) | 0 | 1
Dental Caries (Gastrointestinal disorders) | 1 | 0
Diaphragmatic Hernia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Enterocolitis Hemorrhage (Gastrointestinal disorders) | 0 | 1
Eosinophilic Colitis (Gastrointestinal disorders) | 1 | 0
Erosive Esophagitis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gallstone Ileus (Gastrointestinal disorders) | 1 | 0
Gastric Polyps (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Gastroduodenal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Ulcer Hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Vascular Malformation (Gastrointestinal disorders) | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1
Ileitis (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia Strangulated (Gastrointestinal disorders) | 1 | 0
Intestinal Hematoma (Gastrointestinal disorders) | 1 | 0
Intestinal Ischemia (Gastrointestinal disorders) | 0 | 1
Intestinal Polyp Hemorrhage (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 1 | 0
Lip Edema (Gastrointestinal disorders) | 0 | 1
Lip Swelling (Gastrointestinal disorders) | 0 | 1
Megacolon (Gastrointestinal disorders) | 1 | 0
Mouth Cyst (Gastrointestinal disorders) | 0 | 1
Esophageal Food Impaction (Gastrointestinal disorders) | 1 | 0
Esophageal Obstruction (Gastrointestinal disorders) | 1 | 0
Esophageal Ulcer (Gastrointestinal disorders) | 0 | 1
Esophagitis Ulcerative (Gastrointestinal disorders) | 1 | 0
Pancreatic Cyst (Gastrointestinal disorders) | 0 | 1
Pancreatic Pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis Chronic (Gastrointestinal disorders) | 1 | 0
Pancreatitis Hemorrhagic (Gastrointestinal disorders) | 1 | 0
Pancreatitis Necrotising (Gastrointestinal disorders) | 1 | 0
Pancreatitis Relapsing (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 1
Polyp Colorectal (Gastrointestinal disorders) | 1 | 0
Retroperitoneal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Tongue Cyst (Gastrointestinal disorders) | 1 | 0
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 0 | 1
Volvulus Of Small Bowel (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 52 | 67
Transient Ischemic Attack (Nervous system disorders) | 16 | 19
Presyncope (Nervous system disorders) | 13 | 8
Dizziness (Nervous system disorders) | 9 | 9
Sciatica (Nervous system disorders) | 7 | 8
Headache (Nervous system disorders) | 5 | 4
Vertibrobasilar Insufficiency (Nervous system disorders) | 5 | 3
Loss Of Consciousness (Nervous system disorders) | 4 | 2
Paresthesia (Nervous system disorders) | 5 | 1
Subarachnoid Hemorrhage (Nervous system disorders) | 4 | 1
Convulsion (Nervous system disorders) | 2 | 2
Amnesia (Nervous system disorders) | 2 | 1
Cerebral Hemorrhage (Nervous system disorders) | 3 | 0
Diabetic Neuropathy (Nervous system disorders) | 0 | 2
Hypoesthesia (Nervous system disorders) | 1 | 1
Lumbar Radiculopathy (Nervous system disorders) | 2 | 0
Migraine (Nervous system disorders) | 2 | 0
Nerve Root Lesion (Nervous system disorders) | 0 | 2
Radial Nerve Palsy (Nervous system disorders) | 1 | 1
Viith Nerve Paralysis (Nervous system disorders) | 1 | 1
Acute Disseminated Encephalomyelitis (Nervous system disorders) | 0 | 1
Altered State of Consciousness (Nervous system disorders) | 1 | 0
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 0 | 1
Carotid Artery Stenosis (Nervous system disorders) | 0 | 1
Carotid Sinus Syndrome (Nervous system disorders) | 1 | 0
Cauda Equina Syndrome (Nervous system disorders) | 0 | 1
Cerebral Arteriosclerosis (Nervous system disorders) | 1 | 0
Cerebral Artery Stenosis (Nervous system disorders) | 1 | 0
Cerebral Cyst (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Cognitive Disorder (Nervous system disorders) | 1 | 0
Complex Partial Seizure (Nervous system disorders) | 0 | 1
Coordination Abnormal (Nervous system disorders) | 1 | 0
Dementia With Lewey Bodies (Nervous system disorders) | 0 | 1
Demyelinating Polyneuropathy (Nervous system disorders) | 0 | 1
Dizziness Exertional (Nervous system disorders) | 1 | 0
Dizziness Postural (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Facial Paresis (Nervous system disorders) | 1 | 0
Guillain-Barre Syndrome (Nervous system disorders) | 1 | 0
Hemorrhage Intracranial (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hypoglycemic Coma (Nervous system disorders) | 0 | 1
Hypoglycemic Unconsciousness (Nervous system disorders) | 1 | 0
Intracranial Aneurysm (Nervous system disorders) | 0 | 1
Meningorrhagia (Nervous system disorders) | 1 | 0
Metabolic Encephalopathy (Nervous system disorders) | 0 | 1
Motor Neuron Disease (Nervous system disorders) | 1 | 0
Multiple Sclerosis (Nervous system disorders) | 0 | 1
Multiple Sclerosis Relapse (Nervous system disorders) | 0 | 1
Myasthenia Gravis (Nervous system disorders) | 0 | 1
Myelitis Transverse (Nervous system disorders) | 0 | 1
Nerve Root Compression (Nervous system disorders) | 0 | 1
Nervous System Disorder (Nervous system disorders) | 0 | 1
Neuritis (Nervous system disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0
Psychomotor Hyperactivity (Nervous system disorders) | 1 | 0
Radicular Syndrome (Nervous system disorders) | 0 | 1
Ruptured Cerebral Aneurysm (Nervous system disorders) | 0 | 1
Senile Dementia (Nervous system disorders) | 0 | 1
Speech Disorder (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0
Toxic Encephalopathy (Nervous system disorders) | 0 | 1
Transient Global Amnesia (Nervous system disorders) | 1 | 0
Trigeminal Neuralgia (Nervous system disorders) | 1 | 0
Vertebral Artery Stenosis (Nervous system disorders) | 0 | 1
Vertigo CNS Origin (Nervous system disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 31 | 32
Intervertebral Disk Protrusion (Musculoskeletal and connective tissue disorders) | 15 | 15
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 20 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 12
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 7 | 6
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 5 | 7
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 2 | 6
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 2
Intervertebral Disk Disorder (Musculoskeletal and connective tissue disorders) | 1 | 3
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Fracture Nonunion (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle Hemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 2
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 1
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Nose Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Sensation Of Heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon Calcification (Musculoskeletal and connective tissue disorders) | 0 | 1
Ulnocarpal Abutment Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 11 | 6
Hip Fracture (Injury, poisoning and procedural complications) | 8 | 7
Post Procedural Hemorrhage (Injury, poisoning and procedural complications) | 8 | 5
Head Injury (Injury, poisoning and procedural complications) | 5 | 6
Femur Fracture (Injury, poisoning and procedural complications) | 7 | 2
Subdural Hematoma (Injury, poisoning and procedural complications) | 3 | 6
Fall (Injury, poisoning and procedural complications) | 6 | 2
Foot Fracture (Injury, poisoning and procedural complications) | 3 | 4
Tibia Fracture (Injury, poisoning and procedural complications) | 2 | 5
Humerus Fracture (Injury, poisoning and procedural complications) | 4 | 2
Lower Limb Fracture (Injury, poisoning and procedural complications) | 2 | 4
Incisional Hernia (Injury, poisoning and procedural complications) | 3 | 2
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 3 | 2
Laceration (Injury, poisoning and procedural complications) | 3 | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 2 | 2
Overdose (Injury, poisoning and procedural complications) | 3 | 1
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 2 | 2
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 3
Radius Fracture (Injury, poisoning and procedural complications) | 2 | 2
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 3
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 | 3
Upper Limb Fracture (Injury, poisoning and procedural complications) | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Muscle Rupture (Injury, poisoning and procedural complications) | 1 | 2
Rib Fracture (Injury, poisoning and procedural complications) | 2 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 3 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 | 1
Comminuted Fracture (Injury, poisoning and procedural complications) | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 2
Extradural Hematoma (Injury, poisoning and procedural complications) | 1 | 1
Eye Injury (Injury, poisoning and procedural complications) | 2 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 2
Fractured Sacrum (Injury, poisoning and procedural complications) | 1 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 2
In-Stent Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 2 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 1 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 2 | 0
Post Procedural Hematoma (Injury, poisoning and procedural complications) | 0 | 2
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 | 2
Skull Fracture (Injury, poisoning and procedural complications) | 2 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 1
Subdural Hemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 1
Traumatic Intracranial Hemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 2
Wound Necrosis (Injury, poisoning and procedural complications) | 0 | 2
Accident At Home (Injury, poisoning and procedural complications) | 0 | 1
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0 | 1
Anemia Postoperative (Injury, poisoning and procedural complications) | 1 | 0
Animal Bite (Injury, poisoning and procedural complications) | 1 | 0
Back Injury (Injury, poisoning and procedural complications) | 0 | 1
Brain Contusion (Injury, poisoning and procedural complications) | 1 | 0
Cardiac Procedure Complication (Injury, poisoning and procedural complications) | 1 | 0
Cartilage Injury (Injury, poisoning and procedural complications) | 0 | 1
Chemical Injury (Injury, poisoning and procedural complications) | 1 | 0
Complications Of Transplanted Heart (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of Vertebra (Injury, poisoning and procedural complications) | 0 | 1
Electric Shock (Injury, poisoning and procedural complications) | 1 | 0
Eye Penetration (Injury, poisoning and procedural complications) | 1 | 0
Face Injury (Injury, poisoning and procedural complications) | 1 | 0
Femoral Nerve Injury (Injury, poisoning and procedural complications) | 1 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign Body (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1 | 0
Incisional Hernia, Obstructive (Injury, poisoning and procedural complications) | 0 | 1
Injury Corneal (Injury, poisoning and procedural complications) | 0 | 1
Jaw Fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0
Limb Crushing Injury (Injury, poisoning and procedural complications) | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 1
Open Wound (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Pulmonary Embolism (Injury, poisoning and procedural complications) | 0 | 1
Post Traumatic Pain (Injury, poisoning and procedural complications) | 0 | 1
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural Hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural Hypotension (Injury, poisoning and procedural complications) | 1 | 0
Procedural Vomiting (Injury, poisoning and procedural complications) | 1 | 0
Scapula Fracture (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Skeletal Injury (Injury, poisoning and procedural complications) | 0 | 1
Skin Injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal Cord Injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal Cord Injury Cervical (Injury, poisoning and procedural complications) | 0 | 1
Sternal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon Injury (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Arthritis (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Arthropathy (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Liver Injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Renal Injury (Injury, poisoning and procedural complications) | 1 | 0
Vascular Pseudoaneurism (Injury, poisoning and procedural complications) | 0 | 1
Wound Secretion (Injury, poisoning and procedural complications) | 1 | 0
Chronic Pulmonary Obstructive Disease (Respiratory, thoracic and mediastinal disorders) | 27 | 21
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 | 15
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 15 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 11
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Esophageal Swelling (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Microemboli (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 31 | 14
Hypotension (Vascular disorders) | 10 | 10
Deep Vein Thrombosis (Vascular disorders) | 11 | 8
Hypertensive Crisis (Vascular disorders) | 9 | 8
Orthostatic Hypotension (Vascular disorders) | 3 | 3
Peripheral Arterial Occlusive Disease (Vascular disorders) | 3 | 3
Accelerated Hypertension (Vascular disorders) | 3 | 1
Hematoma (Vascular disorders) | 2 | 2
Thrombophlebitis (Vascular disorders) | 1 | 3
Aortic Aneurism (Vascular disorders) | 2 | 1
Varicose Vein (Vascular disorders) | 3 | 0
Thrombosis (Vascular disorders) | 1 | 1
Aortic Aneurism Rupture (Vascular disorders) | 1 | 0
Aortic Atherosclerosis (Vascular disorders) | 0 | 1
Arterial Hemorrhage (Vascular disorders) | 1 | 0
Arterial Rupture (Vascular disorders) | 1 | 0
Arterial Thrombosis Limb (Vascular disorders) | 0 | 1
Blood Pressure Inadequately Controlled (Vascular disorders) | 0 | 1
Circulatory Collapse (Vascular disorders) | 0 | 1
Diabetic Vascular Disorder (Vascular disorders) | 0 | 1
Endothelial Dysfunction (Vascular disorders) | 1 | 0
Femoral Arterial Stenosis (Vascular disorders) | 1 | 0
Hemorrhage (Vascular disorders) | 0 | 1
Hyperemia (Vascular disorders) | 0 | 1
Hypovolemic Shock (Vascular disorders) | 0 | 1
Labile Hypertension (Vascular disorders) | 1 | 0
Malignant Hypertension (Vascular disorders) | 0 | 1
Popliteal Artery Entrapment (Vascular disorders) | 0 | 1
Shock Hemorrhage (Vascular disorders) | 0 | 1
Venus Insufficiency (Vascular disorders) | 0 | 1
Venus Thrombosis Limb (Vascular disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 17 | 19
Nephrolithiasis (Renal and urinary disorders) | 8 | 11
Calculus Ureteric (Renal and urinary disorders) | 6 | 6
Renal Colic (Renal and urinary disorders) | 4 | 8
Renal Failure (Renal and urinary disorders) | 7 | 5
Hematuria (Renal and urinary disorders) | 5 | 4
Acute Prerenal Failure (Renal and urinary disorders) | 2 | 5
Renal Failure Chronic (Renal and urinary disorders) | 2 | 2
Urinary Retention (Renal and urinary disorders) | 3 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 2
Tubulointerstitial Nephritis (Renal and urinary disorders) | 2 | 1
Urethral Stenosis (Renal and urinary disorders) | 1 | 2
Calculus Bladder (Renal and urinary disorders) | 2 | 0
Hemorrhage Urinary Tract (Renal and urinary disorders) | 1 | 1
Postrenal Failure (Renal and urinary disorders) | 0 | 2
Renal Hemorrhage (Renal and urinary disorders) | 1 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 2
Ureteric Stenosis (Renal and urinary disorders) | 1 | 1
Bladder Fibrosis (Renal and urinary disorders) | 1 | 0
Bladder Neck Obstruction (Renal and urinary disorders) | 1 | 0
Bladder Neck Stenosis (Renal and urinary disorders) | 0 | 1
Bladder Stenosis (Renal and urinary disorders) | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 1 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 1
Obstructive Uropathy (Renal and urinary disorders) | 0 | 1
Pelvic-Ureteric Obstruction (Renal and urinary disorders) | 0 | 1
Renal Mass (Renal and urinary disorders) | 1 | 0
Stag Horn Calculus (Renal and urinary disorders) | 1 | 0
Ureteric Obstructive (Renal and urinary disorders) | 1 | 0
Urethral Pain (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 14 | 16
Cholecystitis Acute (Hepatobiliary disorders) | 10 | 14
Cholecystitis (Hepatobiliary disorders) | 8 | 10
Bile Duct Stone (Hepatobiliary disorders) | 1 | 3
Cholangitis (Hepatobiliary disorders) | 3 | 1
Hepatic Cirrhosis (Hepatobiliary disorders) | 4 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 2 | 1
Biliary Colic (Hepatobiliary disorders) | 0 | 2
Drug Induced Liver Injury (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Jaundice Cholestatic (Hepatobiliary disorders) | 1 | 0
Porcelain Gallbladder (Hepatobiliary disorders) | 0 | 1
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 6 | 8
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 4 | 9
Hypoglycemia (Metabolism and nutrition disorders) | 8 | 5
Dehydration (Metabolism and nutrition disorders) | 7 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 5
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 3 | 2
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetic Complication (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 8 | 8
Anxiety (Psychiatric disorders) | 1 | 5
Confusional State (Psychiatric disorders) | 4 | 2
Major Depression (Psychiatric disorders) | 4 | 2
Suicide Attempt (Psychiatric disorders) | 1 | 5
Mental Status Change (Psychiatric disorders) | 2 | 3
Suicidal Ideation (Psychiatric disorders) | 1 | 3
Completed Suicide (Psychiatric disorders) | 1 | 2
Personality Disorder (Psychiatric disorders) | 0 | 2
Abnormal Behavior (Psychiatric disorders) | 0 | 1
Adjustment Disorder (Psychiatric disorders) | 0 | 1
Alcohol Abuse (Psychiatric disorders) | 1 | 0
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 | 0
Anxiety Disorder (Psychiatric disorders) | 0 | 1
Bipolar Disorder (Psychiatric disorders) | 0 | 1
Bipolar I Disorder (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Delirium Tremens (Psychiatric disorders) | 1 | 0
Depression Suicidal (Psychiatric disorders) | 1 | 0
Disorientaion (Psychiatric disorders) | 0 | 1
Panic Disorder With Agoraphobia (Psychiatric disorders) | 0 | 1
Panic Action (Psychiatric disorders) | 1 | 0
Schizoaffective Disorder (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 2
Hemorrhagic Anemia (Blood and lymphatic system disorders) | 0 | 2
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Acquired Hemophilia (Blood and lymphatic system disorders) | 0 | 1
Anemia Hemolytic Autoimmune (Blood and lymphatic system disorders) | 0 | 1
Deficiency Anemia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Hypochromic Anemia (Blood and lymphatic system disorders) | 0 | 1
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Microcytic Anemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Normochromic Normocytic Anemia (Blood and lymphatic system disorders) | 0 | 1
Splenic Hemorrhage (Blood and lymphatic system disorders) | 1 | 0
Spontaneous Hemotoma (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 9 | 8
Prostatitis (Reproductive system and breast disorders) | 3 | 2
Epididymitis (Reproductive system and breast disorders) | 2 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 1
Uterine Prolapse (Reproductive system and breast disorders) | 1 | 1
Breast Disorder (Reproductive system and breast disorders) | 1 | 0
Breast Pain (Reproductive system and breast disorders) | 1 | 0
Cervical Polyp (Reproductive system and breast disorders) | 1 | 0
Erectile Disfunction (Reproductive system and breast disorders) | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0
Ovarian Cyst Torsion (Reproductive system and breast disorders) | 1 | 0
Pelvic Floor Muscle Weakness (Reproductive system and breast disorders) | 1 | 0
Postmenopausal Hemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatic Obstruction (Reproductive system and breast disorders) | 1 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Rectocele (Reproductive system and breast disorders) | 1 | 0
Spermatocele (Reproductive system and breast disorders) | 1 | 0
Uterine Hemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine Polyp (Reproductive system and breast disorders) | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 3
Arteriogram Coronary (Investigations) | 1 | 1
Blood Pressure Increase (Investigations) | 2 | 0
Cardiac Stress Test Abnormal (Investigations) | 1 | 1
Ejection Fraction Decreased (Investigations) | 1 | 1
Exercise Test Abnormal (Investigations) | 1 | 1
International Normalized Ratio Increased (Investigations) | 1 | 1
Blood Glucose Increased (Investigations) | 1 | 0
Blood Pressure Abnormal (Investigations) | 0 | 1
Echocardiogram Abnormal (Investigations) | 0 | 1
Hemoglobin Decreased (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0
International Normalized Ratio Abnormal (Investigations) | 1 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 1
Pulse Absent (Investigations) | 0 | 1
Urine Output Increased (Investigations) | 0 | 1
Weight Decreased (Investigations) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 5 | 5
Hypoacusis (Ear and labyrinth disorders) | 2 | 1
Vertigo Positional (Ear and labyrinth disorders) | 0 | 3
Deafness Unilateral (Ear and labyrinth disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Meniere's Disease (Ear and labyrinth disorders) | 0 | 1
Sudden Loss Of Hearing (Ear and labyrinth disorders) | 0 | 1
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 | 1
Vestibular Disorder (Ear and labyrinth disorders) | 0 | 1
Leukocytoclastic Vasculitis (Skin and subcutaneous tissue disorders) | 1 | 2
Skin Ulcer (Skin and subcutaneous tissue disorders) | 3 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Bulbous (Skin and subcutaneous tissue disorders) | 0 | 1
Digital Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing Nails (Skin and subcutaneous tissue disorders) | 1 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 1 | 0
Neuropathic Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 4
Anaphylactic Shock (Immune system disorders) | 3 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 2
Antiphospholipid Syndrome (Immune system disorders) | 1 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 1
Allergy For Arthropod Bite (Immune system disorders) | 0 | 1
Amyloidosis (Immune system disorders) | 1 | 0
Multiple Allergies (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1
Hydrocele (Immune system disorders) | 0 | 2
Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 | 0
Atrial Septal Defect (Congenital, familial and genetic disorders) | 0 | 1
Gastrointestinal Arteriovenous Malformation (Congenital, familial and genetic disorders) | 0 | 1
Hemorrhagic Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 | 0
Keratosis Folicular (Congenital, familial and genetic disorders) | 0 | 1
Laryngocele (Congenital, familial and genetic disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 2
Hypercalcemia of Malignancy (Endocrine disorders) | 1 | 0
Hyperparathyroidism (Congenital, familial and genetic disorders) | 0 | 1
Hypopituitarism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Carcinoma Basocellular (Noze) (General disorders) | 0 | 1 — Body System Not Defined
Contusion Left Knee (General disorders) | 1 | 0 — Body System Not Defined
Dislodgment Of Gastronomy Tube (General disorders) | 1 | 0 — Body System Not Defined
Gastrointestinal Stomal Tumor (General disorders) | 0 | 1 — Body System Not Defined
Sigmoid Colon Adenocarcinoma (General disorders) | 1 | 0 — Body System Not Defined
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dalcetrapib (RO4607381) (N=7938) | Placebo (N=7933)
Nasopharyngitis (Infections and infestations) | 438 | 460
Chest Pain (General disorders) | 833 | 830
Fatigue (General disorders) | 396 | 416
Edema Peripheral (General disorders) | 300 | 393
Diarrhea (Gastrointestinal disorders) | 541 | 342
Angina Pectoris (Cardiac disorders) | 585 | 569
Cough (Respiratory, thoracic and mediastinal disorders) | 403 | 415
Dizziness (Nervous system disorders) | 413 | 459
Hypertension (Vascular disorders) | 578 | 513

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No